CLINICAL TRIAL: NCT06243549
Title: Exploring the Associations Between the Biomechanical and Psychological Mechanistic Pathways of Lower Back Pain Development Amongst Persons With Lower-Limb Amputation
Brief Title: Personalisation of Prosthetic Care for Lower- Limb Amputees
Status: Active, not recruiting | Type: Observational
Sponsor: University of Bath (Other)
Collaborators: University Hospitals Bristol and Weston NHS Foundation Trust (Other); Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Principal Investigator, Alexandra Withey, Principal Investigator, University of Bath
Other Study IDs: 321729
Record Dates: First submitted 2024-01-25; First posted 2024-02-06 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The global rise in lower-limb amputations is mainly due to diabetes and vascular complications. Amputations cause serious physical and psycho-social disabilities which impair locomotion and compromise patients quality of life. Biopsychosocial factors such as altered gait parameters, poor prosthetic fit, depression, fear avoidance behaviours and stigma increase the risk of individuals incurring lower back pain; the leading cause of secondary disability amongst persons with lower-limb amputation. Exploring the potential mechanistic pathways of lower back pain development is important to inform timely patient-centred programmes of care. Currently, limited information exists to inform the design of such programmes. Thus, there is a pressing need to understand the bio-behavioural, psychological, and social features of individuals with lower-limb amputation in the presence of lower back pain.

DETAILED DESCRIPTION:
Studies yield conclusive findings on the biomechanical characteristics of the gait of persons with lower-limb amputation wearing a prosthetic limb, however there are discrepancies between the variables analysed by different studies and the parameters that may predict the development of secondary pain conditions, such as lower back pain, knee osteoarthritis and osteoporosis and best functional outcomes are unknown.

Lower back pain and joint pain can be a symptom of musculoskeletal diseases among persons with lower-limb amputation and can influence one's gait and functional outcomes. Although the association between lower-limb amputation and lower back pain is clear, understanding the timings, the propagators and mechanisms related to lower back pain among persons with lower-limb amputation is important to inform care management and rehabilitation programmes. Currently, there is a gap in the literature regarding the role of key determinants on functional outcomes among persons with lower-limb amputation and when they start appearing. Also, it is not clear what is the association between biomechanical gait parameters, muscle activations and pain. Further multidisciplinary research is required to investigate the relationship between different forms of pain among persons with lower-limb amputation and biomechanical gait variables, and how these change over time. This knowledge can then be used to form a prognosis of functional outcomes among persons with lower-limb amputation and appropriate rehabilitation programmes can be developed for different populations of amputations.

This project aims to identify the determinants of lower back pain among persons with unilateral lower-limb amputation, over a period of 12-months after their amputation. Additionally, the relationships between gait characteristics, trunk and lower-limb muscle activations and different sources of pain will be investigated. This information will be used to identify the predictive characteristics of the musculoskeletal diseases, such as lower back pain, and will inform future care management and rehabilitation processes.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Unilaterally amputated
* Able to walk on level ground
* Newly fitted with a prosthetic (0-3-months post-amputation)

Exclusion Criteria:

* Balance disorders
* Patients who lack the capacity to consent for prosthetic use
* Patients at serious risk of sound foot which limits normal rehabilitation
* Transfer-in patients
* Persons with congenital lower-limb amputation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment of persons with unilateral TFA and TTA of both vascular and traumatic aetiology will be attempted from the Bristol Centre for Enablement and the Portsmouth Enablement Centre (North Bristol NHS Trust and Portsmouth Hospitals University NHS Trust, respectively).
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
How do gait characteristics and muscle activations influence functional outcomes post-amputation and how do these variables influence the development of lower back pain? | 12-months
  Monitoring patients gait and muscle activities of the erector spinae, latissimus dorsi, gluteus medius, and sound limb biceps femoris and rectus femoris, during walking at self-selected speed, and how these variables influence lower back pain, assessed through the Roland-Morris Disability Questionnaire (no scale, greater number of statements circled indicates a worse outcome; maximum score of 24), and patient functional outcomes, where the term 'function' refers to the comprehensive overview of each participant's everyday interactions and long-term targets, defined by the participant in terms of person-specific activities and goals.

SECONDARY OUTCOMES:
How does the gait of persons with lower-limb loss change over a period of 12-months? | 12-months
  Monitoring patients gait during walking at self-selected speed over a period of 12-months. Key outcomes measures include lower-limb and lumbar kinetics (e.g., joint reaction forces), lower-limb kinematics, including lumbopelvic and lower-limb region movement asymmetries (e.g., joint angles), body centre of mass position and symmetry indices, and temporal-spatial characteristics of gait (e.g., stride frequency, walking speed).
What is the time-scale for the development of lower back pain post-amputation? | 12-months
  Looking at the time-scale for the development of lower back pain, assessed using online questionnaires, over a period of 12-months. The online questionnaires include the Brief Pain Inventory (scale of 0-10; higher score = worse outcome), Pain Catastrophising Scale (scale of 0-4; higher score = worse outcome), Tampa Scale for Kinesiophobia (scale of 1-4; higher score = worse outcome), the Roland-Morris Disability Questionnaire (no scale, greater number of statements circled indicates a worse outcome; maximum score of 24), State Trait Anxiety Index Y form (scale of 1-4; higher score = worse outcome), Patient Health Questionnaire (scale of 0-3; higher score = worse outcome), Short Form 36 Health Survey Questionnaire (scale of 1-3; higher score = better outcomes), and the International Physical Activity Questionnaire (no scale, patients indicate the number of hours spent per day doing different activities such as walking).
What is the relationship between lower back pain and other types of pain? | 12-months
  Looking at the relationship between lower back pain and other types of pain, including joint pain, phantom limb pain, residual limb pain. Pain will be assessed through online questionnaires.
  The online questionnaires include the Brief Pain Inventory (scale of 0-10; higher score = worse outcome), Pain Catastrophising Scale (scale of 0-4; higher score = worse outcome), Tampa Scale for Kinesiophobia (scale of 1-4; higher score = worse outcome), the Roland-Morris Disability Questionnaire (no scale, greater number of statements circled indicates a worse outcome; maximum score of 24), State Trait Anxiety Index Y form (scale of 1-4; higher score = worse outcome), Patient Health Questionnaire (scale of 0-3; higher score = worse outcome), Short Form 36 Health Survey Questionnaire (scale of 1-3; higher score = better outcomes), and the International Physical Activity Questionnaire (no scale, patients indicate the number of hours spent per day doing different activities such as walking).
How many persons with lower-limb amputation develop lower back pain over the 12-month monitoring period? | 12-months
  The research question aims to quantifying the incidence of lower back pain development amongst the population of persons with unilateral lower limb amputation included in the study.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Bristol Centre for Enablement, Bristol
  - Portsmouth Enablement Centre, Portsmouth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Withey A, Cazzola D, Tabor A, Seminati E. Exploring the associations between the biomechanical and psychological mechanistic pathways of lower back pain development amongst persons with lower-limb amputation: A study protocol. PLoS One. 2025 Feb 6;20(2):e0314523. doi: 10.1371/journal.pone.0314523. eCollection 2025. PMID 39913459